CLINICAL TRIAL: NCT07226544
Title: A Phase II Study of Neoadjuvant Ivonescimab in Patients With High-Risk, Localized RCC
Brief Title: Ivonescimab Prior to Surgery for the Treatment of High-Risk Localized Clear Cell Renal Cell Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25395; NCI-2025-07733 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25395 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Localized Clear Cell Renal Cell Carcinoma; Resectable Clear Cell Renal Cell Carcinoma; Stage II Renal Cell Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Biopsy; Specimen Handling; Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ivonescimab) (Experimental): Patients receive ivonescimab IV over 60-120 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Between 4-10 weeks after completion of ivonescimab treatment, patients then undergo SOC nephrectomy. Patients also undergo ECHO during screening, biopsy prior to treatment start, and CT and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Ivonescimab; Procedure: Nephrectomy; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Ivonescimab — Given IV
  Other Names: AK 112; AK-112; AK112; Anti-PD-1/Anti-VEGF Bispecific Antibody AK112; Anti-PD-1/VEGF Bispecific Antibody AK112; PD-1/VEGF Bispecific Antibody AK112; SMT 112; SMT-112; SMT112
Procedure: Nephrectomy — Undergo SOC nephrectomy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well ivonescimab works prior to surgery in treating patients with high-risk clear cell kidney (renal cell) cancer that has not spread to other parts of the body (localized). Immunotherapy with monoclonal antibodies, such as ivonescimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ivonescimab may also stop or slow the cancer by blocking the growth of new blood vessels necessary for tumor growth. Giving ivonescimab before standard surgery may make the tumor smaller.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the response rate associated with ivonescimab in patients with high-risk, localized renal cell carcinoma (RCC) planned for nephrectomy.

SECONDARY OBJECTIVES:

I. To define toxicity associated with ivonescimab in this setting. II. To define the feasibility of surgery following systemic therapy with ivonescimab.

III. To determine the pathologic response rate following ivonescimab. IV. To characterize KIM-1 expression before and after ivonescimab. V. To determine survival outcomes following ivonescimab.

EXPLORATORY OBJECTIVES:

I. To characterize the expression of validated genomic signatures (including those derived from IMmotion151) in baseline biopsy and nephrectomy tissue (i.e., before and after therapy with ivonescimab).

II. To evaluate patient-reported quality of life using the FKSI-23 instrument at baseline, pre-surgery, and at post-surgical follow-up time points.

OUTLINE:

Patients receive ivonescimab intravenously (IV) over 60-120 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for 4 cycles in the absence of disease progression or unacceptable toxicity. Between 4-10 weeks after completion of ivonescimab treatment, patients then undergo standard of care (SOC) nephrectomy. Patients also undergo echocardiogram (ECHO) during screening, biopsy prior to treatment start, and computed tomography (CT) and blood sample collection throughout the study.

After completion of study treatment, patients are followed every 12 weeks for a total of 2 years and then periodically at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of clear cell RCC
* High-risk disease defined as cT2G3-4N0M0, cT3GanyN0M0, cT4GanyN0M0, cTanyGanyN+M0 (Grade determined by biopsy)
* Candidate for partial or complete nephrectomy that extirpates all tumor tissue as part of treatment plan
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (no blood transfusions or growth factor therapy used within 7 days of the screening complete blood count [CBC])
* Platelet count ≥ 100 × 10^9/L (no blood transfusions or growth factor therapy used within 7 days of the screening CBC)
* Hemoglobin ≥ 9.0 g/dL (no blood transfusions or growth factor therapy used within 7 days of the screening CBC)
* Creatinine clearance (CrCL) ≥ 50 mL/min using the Cockcroft-Gault formula or estimated glomerular filtration rate (eGFR) value ≥ 60 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (adjustment by body surface area [BSA] is not required for eGFR)
* Urine protein < 2+ or 24-hour urine protein quantification < 1.0 g
* Serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); For patients with liver metastases or confirmed/suspected Gilbert syndrome, TBIL ≤ 3 × ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; For patients with liver metastases, AST and ALT ≤ 5 × ULN
* Coagulation: Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 × ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy). This applies only to patients who are not on therapeutic anti-coagulation. Patients receiving therapeutic anti-coagulation should be on a stable dose
* Female patients of childbearing age must have negative serum pregnancy test results before enrollment or per region-specific guidance documented in the informed consent and a negative urine pregnancy test on the day of first dose prior to dosing
* Female patient of childbearing potential having sex with an unsterilized male partner must agree to use a highly effective method of contraception from the beginning of screening until 90 days after the last dose of the ivonescimab
* Unsterilized male patients having sex with a female partner of childbearing potential, or a pregnant or breastfeeding partner must agree to use barrier contraception (male condom) for the duration of the treatment period until 90 days after the last dose of ivonescimab. Male patients with female partners of childbearing potential must have the female partner agree to use at least 1 form of highly effective contraception for the duration of the treatment period until 90 days after the last dose of ivonescimab
* Adults aged 18 years or older

Exclusion Criteria:

* Prior systemic anti-tumor treatment for RCC
* Major surgical procedures or serious trauma within 4 weeks prior to enrollment, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to enrollment
* History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to enrollment, including but not limited to:

  * Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to enrollment is not allowed. The use of full-dose anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits according to the medical standard of the enrolling institution
* Poorly controlled hypertension with repeated systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy
* Active autoimmune or lung disease requiring systemic therapy (eg, with disease modifying drugs, prednisone > 10 mg daily or equivalent, immunosuppressant therapy) within 2 years prior to enrollment, however the following will be allowed:

  * Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted
  * Intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections is permitted
* History of major diseases before enrollment, specifically:

  * Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or unstable vascular disease (eg, aortic aneurysm at risk of rupture, Moyamoya disease) that required hospitalization within 12 months prior to enrollment, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
  * History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before enrollment
  * History of any grade arterial thromboembolic event, Grade 3 and above venous thromboembolic event, as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 12 months prior to enrollment
  * Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before enrollment
  * History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to enrollment
* Imaging during the screening period shows that the patient has metastatic disease
* Symptomatic central nervous system (CNS) metastases, CNS metastases with hemorrhagic features, CNS metastasis ≥ 1.5 cm, CNS radiation within 7 days prior to enrolment, potential need for CNS radiation within the first cycle, or leptomeningeal disease
* Live vaccine or live attenuated vaccine within 4 weeks prior to planned enrolment, or if scheduled to receive a live vaccine or live attenuated vaccine during the study period. Inactivated vaccines are permitted
* Severe infection within 4 weeks prior to enrolment, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; active infection (as determined by the investigator) requiring systemic anti-infective therapy within 2 weeks prior to enrolment (excluding antiviral therapy for hepatitis B or C)
* Has pre-existing peripheral neuropathy that is ≥ Grade 2 by CTCAE version 5
* Uncontrolled pleural effusions, pericardial effusions, or ascites that is clinically symptomatic
* History of non-infectious pneumonia requiring systemic corticosteroids, or current interstitial lung disease
* Active or prior history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Known history of human immunodeficiency virus (HIV) whose viral load is not controlled
* Current use of systemic corticosteroids (> 10 mg daily prednisone or equivalent)
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Patients with active hepatitis B are required to have stable or declining levels of hepatitis B DNA by polymerase chain reaction (PCR) on appropriate anti-viral therapy with acceptable tolerability for one month prior to enrolment. All patients with active hepatitis C (hepatitis C virus [HCV] antibody positive with HCV ribonucleic acid [RNA] levels above the lower limit of detection) are excluded
* Known allergy to any component of any study drug; known history of severe hypersensitivity to other monoclonal antibodies
* History or current evidence of any condition (medical [including adverse events from prior anticancer therapy, disorders secondary to tumor], surgical or psychiatric [including substance abuse]), or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, might lead to higher medical risk and/or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Patient is breastfeeding or plans to breastfeed during the study
* History of severe immune-mediated adverse events from immunotherapy agents (i.e. PD1/PDL1/CTLA4 inhibitors), or immune-related ocular toxicity, pneumonitis, or cardiomyopathy of any grade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-06-08 (Estimated); Primary Completion 2027-09-08 (Estimated); Study Completion 2027-09-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a best overall response (ORR) | Up to 2 years after completion of study treatment
  Objective response is defined as complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors. The ORR will be estimated as the proportion of patients who have CR or PR during the treatment, along with the 90% and 95% exact confidence intervals.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after completion of study treatment
  Will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5.0. Safety and toxicity will be assessed by tabulating the toxicity type, frequency, grades and proportion identified in the participants treated on the trial. Binary proportions and associated confidence intervals will be calculated.
Rate of completion of surgery | At least 4 weeks after and within 10 weeks of the last cycle of ivonescimab (each cycle is 21 days)
  Proportion of patients who undergo the planned nephrectomy
Pathologic complete response (pCR) | Up to 2 years after completion of study treatment
  pCR defined as 0% viable tumor cells in the nephrectomy specimen and sampled regional lymph nodes at the time of surgery, assessed per NCI standards and confirmed by central pathology review. The pCR rate will be estimated as the proportion of all treated patients who undergo surgery and have pCR; patients who do not undergo surgery or have an unevaluable specimen will be considered non-responders. Will be estimated as the proportion of patients who have CR, major response, or PR, after the treatment, along with confidence intervals.
Peri-treatment KIM-1 levels | Prior to surgery and after completion of Cycle 4 (each cycle is 21 days)
  Stored plasma will be analyzed for KIM-1 and other exploratory analytes.
Recurrence-free survival | From date of surgery to disease recurrence or death from any cause, whichever occurs first, assessed up to 2 years after completion of study treatment
  The method of Kaplan-Meier will be used to estimate survival distributions.
Overall survival | From the start of study therapy to death from any cause, assessed up to 2 years after completion of study treatment
  The method of Kaplan-Meier will be used to estimate survival distributions.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Yip, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States